CLINICAL TRIAL: NCT02071264
Title: Effects of an HIV Intervention Among Female and Male Entertainers and Spa/Sauna Workers in the Philippines
Brief Title: Effects of an HIV Intervention Among Sex Workers in the Philippines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lianne Urada (Other)
Collaborators: University of California, Los Angeles (Other); Center for Environment and Sustainable Development Foundation, Inc. (Industry); National Institute on Drug Abuse (NIDA) (NIH); The Fordham University HIV and Drug Abuse Prevention Research Ethics Training Institute (RETI) (Other); University of California, San Diego (Other); San Diego State University (Other)
Responsible Party: Sponsor-Investigator, Lianne Urada, Assistant Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Philstudy
Record Dates: First submitted 2014-02-23; First posted 2014-02-25 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: HIV/AIDS Prevention
Keywords: HIV/AIDS; sex work; reproductive health; human rights; ethics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sex Work

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIV/STI intervention (Other): This study implements a socio-behavioral intervention in Metro Manila, the Philippines, using a community-based participatory approach with 1-2 psychosocial and health education training workshops for the establishment managers and their workers, including street sex workers, focusing on HIV/AIDS risk reduction information, condom use, and condom negotiation skill-building. Participants participate in dream-building activities to explore personal goals and goals for their organization of peers. The interventions are directed at organizational behavior change and social influence modeling through training peers and managers. The participants receive information on STIs along with standard care, held on a day convenient to the participants and at a neutral location.
  Interventions: Behavioral: HIV/STI intervention

INTERVENTIONS:
Behavioral: HIV/STI intervention — The intervention covers HIV101 information, reproductive health and human rights national policies, goal setting activities as individuals and as a group, results of prior research on ethics of doing research with sex workers.

SUMMARY:
This study will implement a socio-behavioral intervention in Quezon City, the Philippines, using a community-based participatory approach. The intervention involves 1-2 psychosocial and health education training workshops for the establishment managers and their workers, focusing on HIV/AIDS risk reduction information and condom use and condom negotiation skill-building. Participants will also be invited to do dream-building activities that explore their personal goals and goals for their organization of peers.

DETAILED DESCRIPTION:
This study will implement a socio-behavioral intervention in Quezon City, the Philippines, using a community-based participatory approach. The intervention involves 1-2 psychosocial and health education training workshops for the establishment managers and their workers, focusing on HIV/AIDS risk reduction information, condom use, and condom negotiation skill-building. Participants will also be invited to do dream-building activities that explore their personal goals and goals for their organization of peers.

The intervention involves targeted and tailored bio-psycho-educational interventions directed at organizational behavior change and social influence modeling through training peers and managers. The intervention site will receive peer and manager trainings consisting of specific information on STIs along with standard care, held on a day convenient to the participants and at the establishment or neutral location.

In addition to quick pre-post tests before and immediately after the intervention, participants will be interviewed 6-12 months after the intervention to evaluate the effects of the intervention on their STI/HIV knowledge, attitudes, beliefs, safer sex practices, and social support.

ELIGIBILITY:
Inclusion Criteria:

* self-identification as conducting sex work or working in a venue where sex work occurs.

Exclusion Criteria:

* those not actively engaging in sex work activities or working in a venue or area where sex work occurs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HIV/STI knowledge | 6 months
  Knowledge of HIV/STI transmission and ways to protect oneself

CONTACTS AND LOCATIONS:
Overall Officials: Lianne A Urada, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Center for Environment and Sustainable Development Foundation, Inc., Manila, Philippines

REFERENCES:
- [Background] Urada LA, Morisky DE, Pimentel-Simbulan N, Silverman JG, Strathdee SA. Condom negotiations among female sex workers in the Philippines: environmental influences. PLoS One. 2012;7(3):e33282. doi: 10.1371/journal.pone.0033282. Epub 2012 Mar 20. PMID 22448241
- [Background] Urada LA, Morisky DE, Hernandez LI, Strathdee SA. Social and structural factors associated with consistent condom use among female entertainment workers trading sex in the Philippines. AIDS Behav. 2013 Feb;17(2):523-35. doi: 10.1007/s10461-011-0113-x. PMID 22223297
- [Background] Urada LA, Strathdee SA, Morisky DE, Schilling RF, Simbulan NP, Estacio LR Jr, Raj A. Sex work and its associations with alcohol and methamphetamine use among female bar and spa workers in the Philippines. Asia Pac J Public Health. 2014 Mar;26(2):138-46. doi: 10.1177/1010539512471969. Epub 2013 Jan 22. PMID 23343641
- [Result] Urada LA, Simmons J, Wong B, Tsuyuki K, Condino-Enrera G, Hernandez LI, Simbulan NP, Raj A. A human rights-focused HIV intervention for sex workers in Metro Manila, Philippines: evaluation of effects in a quantitative pilot study. Int J Public Health. 2016 Nov;61(8):945-957. doi: 10.1007/s00038-016-0875-z. Epub 2016 Sep 6. PMID 27600733